CLINICAL TRIAL: NCT02883790
Title: Multicenter, Randomized, Double-blind, Parallel-group, Placebo Controlled, Study to Evaluate the Effects of Melatonin (Somnage®- Food Supplement) in the Management on Sleep Quality and Mood Alteration in Cancer Patients
Brief Title: Effects of Somnage® in the Management on Sleep and Mood in Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrolment rate
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HF02-13-42
Record Dates: First submitted 2016-01-26; First posted 2016-08-30 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2016-08

CONDITIONS: Breast Cancer; Lung Cancer; Colon Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Somnage (Experimental): Group A-Melatonin 1mg, Zinc, Magnesium Oral administration o.d.
  Interventions: Dietary Supplement: Somnage
- Placebo (Placebo Comparator): Oral administration o.d.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Somnage — Melatonin 1mg, Zinc, Magnesium
  Arms: Somnage
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this placebo-controlled randomized study is to evaluate the effects of Melatonin 1mg/Zn 30% VNR/Mg 100% VNR (food supplement) in the management on sleep quality and mood alteration in cancer patients

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the activity of a food supplement, made of Melatonin, Zinc and Magnesium on sleep quality in cancer patients, compared to placebo.

Secondary objectives are to evaluate the activity of Melatonin, Zinc and Magnesium on the quality of life, on the fatigue and on the mood alteration in cancer patients.

The study will also assess the safety of the food supplement under investigation.

In two small subgroups, on voluntary basis, some additional assessments will be done (arm band, nutritional change diary, DXA in one group and activity tracker in another group)

ELIGIBILITY:
Inclusion Criteria:

1. Male and Females aged between 18 and 75 years (included)
2. Pittsburgh Sleep Quality Index (PSQI) score ≥ 5
3. Diagnosed for breast, lung or colon-rectal cancer
4. Metastatic first chemotherapy line
5. Planned duration of chemotherapy treatment at least 63 days
6. Negative to pregnancy test
7. Patients able to swallow

Exclusion Criteria:

1. Known hypersensitivity reaction to Melatonin, Zinc or Magnesium or any components of the product
2. Known current drug or alcohol abuse.
3. Use of other investigational drug(s) within 30 days before study entry or during the study
4. Clinically significant findings on physical examination or presence of known clinically significant disease that would interfere with study evaluation
5. Patients treated with benzodiazepines, hypnotic, anticonvulsant, antipsychotic or antidepressant drugs in the two months before screening visit
6. Patients receiving or planned to receive warfarin
7. Chronic treatment with steroids with daily dose over 10 mg prednisone or equivalent product
8. Brain metastases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-10; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Quality of sleep assessed using the PSQI scale | up to 63 days of treatment
  PSQI scale

SECONDARY OUTCOMES:
Subjective sleep quality through sleep diary | up to 63 days of treatment
  Sleep diary analysis
Overall fatigue assessed using the Brief Fatigue Inventory (BFI) questionnaire | up to 63 days of treatment
  Fatigue assessment through Brief Fatigue Inventory (BFI) questionnaire
Quality of Life evaluated according to SF-12 scale | up to 63 days of treatment
  Quality of Life evaluated according to SF-12 scale

OTHER OUTCOMES:
Number and typology of adverse events | up to 63 days of treatment
  Number and typology of adverse events (AEs), Physical examination, Vital signs, Laboratory tests (hematology, blood chemistry)

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Istituto Nazionale dei Tumori di Milano, Milan
  - I.E.O. Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera S. Gerardo di Monza, Monza
  - Policlinico S. Matteo di Pavia, Pavia
  - Azienda di Servizi alla Persona di Pavia, Pavia

IPD SHARING:
Plan to Share IPD: No